CLINICAL TRIAL: NCT03241030
Title: Sucralfate to Improve Oral Intake in Children With Infectious Oral Ulcers: a Randomized, Double-blind, Placebo-Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Nidhi Vaidya, Resident, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017-06-0024
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Herpangina; Gingivostomatitis; Hand, Foot and Mouth Disease
MeSH Terms: conditions — Herpangina; Hand, Foot and Mouth Disease | interventions — Sucralfate; Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Subjects will receive sucralfate
  Interventions: Drug: Sucralfate; Drug: Acetaminophen; Drug: Ibuprofen
- Placebo Group (Placebo Comparator): Subjects will receive a placebo
  Interventions: Other: Placebo; Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Sucralfate — Will receive 20mg/kg/dose up to 1 gram.
  Arms: Experimental Group
Other: Placebo — Will received placebo solution of similar quantity to that of the weight based dose of sucralfate.
  Arms: Placebo Group
Drug: Acetaminophen — All patients will receive analgesia, either acetaminophen 15mg/kg or ibuprofen 10mg/kg depending on medication administration prior to arrival in the Emergency Department and at the discretion of the treating physician, in addition to either the experimental drug or placebo.
Drug: Ibuprofen — All patients will receive analgesia, either acetaminophen 15mg/kg or ibuprofen 10mg/kg depending on medication administration prior to arrival in the Emergency Department and at the discretion of the treating physician, in addition to either the experimental drug or placebo.

SUMMARY:
The purpose of this study is to see if sucralfate, a medication commonly used for patients with stomach ulcers, may help pediatric patients with mouth ulcers decrease their pain level and improve their ability to drink.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥6 months and ≤5 years old
* Present with oral infectious ulcers such as gingivostomatitis, herpangina, or hand, foot and mouth disease
* History of decreased oral fluid intake by parent or guardian
* English or Spanish speaking parents or guardians

Exclusion Criteria:

* Severely dehydrated or toxic, requiring immediate resuscitation
* Exclusively breastfed
* Severe dental disease
* Significant mouth trauma
* Active Malignancy
* Preexisting upper airway obstruction or swallowing difficulties
* Received intravenous fluids within 24 hours
* Administration of BOTH acetaminophen AND ibuprofen prior to triage and within 4 hours of enrollment

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Vaidya, MD, Principal Investigator — UT Dell Medical School
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh NV, Gabriele GA, Wilkinson MH. Sucralfate as an Adjunct to Analgesia to Improve Oral Intake in Children With Infectious Oral Ulcers: A Randomized, Double-Blind, Placebo-Controlled Trial. Ann Emerg Med. 2021 Sep;78(3):331-339. doi: 10.1016/j.annemergmed.2021.01.019. Epub 2021 Apr 16. PMID 33867179

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Placebo Group
Started | 50 | 52
Completed | 49 | 51
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Placebo Group | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 51 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 24 | 23 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 39 | 42 | 81
  White | 9 | 5 | 14
  African American/Black | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Oral Intake in ml/kg
Description: Will quantify the amount (in ml/kg) of liquid ingested after intervention.
Time Frame: Approximately 60 minutes after medication administration.
Measure: Median (Inter-Quartile Range); unit: oral intake in ml/kg
Arm/Group | Experimental Group | Placebo Group
Number analyzed (Participants) | 49 | 51
oral intake in ml/kg | 9.7 [3.9 to 19.4] | 10.7 [7.2 to 17.1]

2. Secondary Outcome: Number of Participants That Require Intravenous Fluid Administration
Description: To explore the difference in the rates of intravenous fluid (IVF) administration in children treated with sucralfate versus placebo.
Time Frame: 6 hours from the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Placebo Group
Number analyzed (Participants) | 49 | 51
Participants | 5 | 1

3. Secondary Outcome: Number of Participants That Require Admission
Description: To explore the difference in the rates admission rates in children treated with sucralfate versus placebo.
Time Frame: 6 hours from the time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Placebo Group
Number analyzed (Participants) | 49 | 51
Participants | 1 | 2

4. Secondary Outcome: Number of Participants With Unscheduled Visits
Description: Will call families to find out about any unscheduled visits.
Time Frame: Approximately 72 hours from ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Placebo Group
Number analyzed (Participants) | 49 | 51
Participants | 4 | 6

ADVERSE EVENTS:
Time Frame: Until discharge from ED (Average time 3.5 hours)
Arm/Group | Experimental Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03241030/Prot_SAP_002.pdf